CLINICAL TRIAL: NCT02094989
Title: Prospective, Observational Controlled Trial to Assess the Statistical and the Visual Accuracy of the Individual VCG-ECG-Transformation in Dependence of Posture
Brief Title: ECG and VCG in Dependence of Body Posture
Acronym: EVER
Status: Completed | Type: Observational
Sponsor: Bern University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Rolf Oberholzer, MD, Bern University of Applied Sciences
Other Study IDs: BFH-001
Record Dates: First submitted 2014-03-19; First posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Heart Disease; Arrhythmia
Keywords: electrocardiogram; vectorcardiogram; telecardiology; linear regression; individual transformation matrix; posture
MeSH Terms: conditions — Coronary Disease; Arrhythmias, Cardiac

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- diagnostic
  Interventions: Other: posture dependence of VCG-ECG-transformation

INTERVENTIONS:
Other: posture dependence of VCG-ECG-transformation

SUMMARY:
The electrocardiogram (ECG) is an important diagnostic procedure in medicine mainly to detect circulation disorders and problems of the spread of the electrical heart impulse. It is frequently the first measure in clinical practice when angina pectoris, acute myocardial infarction or an arrhythmia are suspected. The ECG is easy to perform, safe and cheap.

Posture changes are known to cause alterations of the ECG [1]. Deviation of the electrical heart axis (EHA) [2], temporary changes of the QRS morphology and ST-segment alterations are of particular importance in view of diagnostic accuracy [3], [4]. In ambulatory ECG recordings ST-segment alterations for instance might mistakenly be interpreted as cardiac ischemia [5]. Artifacts could be minimized by the concurrent determination of the deviation of the electrical heart axis [6] [7]or by using posture detectors [8] helping to correlate ECG changes to posture changes.

Due to the emergence of new computer based opportunities ambulatory ECG in the sense of home monitoring is an emerging market. Together with the superiority compared to the scalar ECG in detecting certain pathologies, like myocardial infarction and right ventricular hypertrophy, the VCG gained new interest in recent years [9]. Four ECG leads are sufficient to synthesize a standard 12-lead ECG from a VCG and vice versa with a transformation matrix [10] [11].The redirection of the spatial VCG after posture changes has been determined for the QRS loop with the Frank leads, which is the reference method for constructing the VCG [12][13].

4 leads of an ambulatory ECG are sufficient to construct the VCG if arranged approximately in the position of three rectangular axes. Doctors are best trained to interpret standard 12 lead ECGs. With optimization of the leads of ambulatory (Holter) ECG towards the three rectangular axes, this might allow mathematical transformation into the standard 12 lead ECG. A precondition would be that the transformation matrix is independent of posture. To date, transformation matrix between Frank VCG and standard 12 lead ECG has only been calculated in resting ECGs [5].

This is the first study which investigates the transformation matrix in different postures. Additionally, the investigators will investigate for the first time prospectively for known artefacts of stress testing and ambulatory ECGs.

Aim:

Simultaneous prospective recording of the standard 12 lead ECG and the Frank-lead VCG in different postures is expected to add information on potential causes of artifacts of the ECG caused by posture changes. During continuous recording, the investigators will investigate the accuracy of the linear affine transformation with posture, the occurrence (dimension and duration) of ECG/ VCG morphology changes and ST-segment alterations, and VCG angle changes in dependence of posture changes in healthy young men.

Hypothesis The investigators hypothesis is that the transformation matrix between Frank-Lead VCG and standard 12-lead ECG is posture dependent.

Artefacts of the ECG due to posture changes are systematic. The knowledge of the systematics improves the diagnostic accuracy of ambulatory ECG and stress testing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects included in the study must meet the following criteria:
* Male aged 18 - 60 years
* Body Mass Index: 18.5 - 35 (WHO: normal weight - overweight - class I obesity)
* Basic pulse rate: 60 - 100 beats per minute
* Blood pressure: max. systolic 140 / diastolic 90 mm Hg

Exclusion Criteria:

* Chronic or acute disease (including drug abuse, bronchial asthma, pulmonary emphysema, COPD)
* Cardiac disease or limitations of the heart function (angina pectoris, previous myocardial infarction, arrhythmia, dyspnea)
* Implants for the treatment of acute and/or chronic diseases
* Regular intake of medication (> 2 per week) for the treatment of acute and/or chronic diseases

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy men without history of cardiac disorder
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
posture dependence of the individual VCG-ECG-Transformation matrix | N/A (one simultaneous ECG/VCG record over 20 minutes)
  The transformation matrix will be defined as independent of posture, if the accuracy between measured and calculated 12 lead ECG of each posture vary below the accuracy level as defined in IEC 60601-1-52.

SECONDARY OUTCOMES:
artifacts in the ECG morphology | N/A (one simultaneous ECG/VCG record over 20 minutes)
  Posture changes will be defined as not being a relevant artifact for QRS morphology- and ST-segment alterations, if the accuracy between the supine standard 12 lead ECG and the measured 12 lead ECG of another posture vary below the accuracy level as defined in IEC 60601-1-52.
posture dependence of electrical heart axis | N/A (one simultaneous ECG/VCG record over 20 minutes)
  The mean, range and standard deviation (SD) of angle changes of the electrical heart axis of each posture of all participants will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- CTU, Bern, Canton of Bern, Switzerland